CLINICAL TRIAL: NCT02881229
Title: Open Ended Chart Review of Adult Women Presenting to the Vulvar Mucosal Specialty Clinic at Northwestern University Department of Dermatology
Brief Title: Vulvar Mucosal Specialty Clinic Chart Review
Status: Terminated | Type: Observational
Why Stopped: Investigator is no longer at Northwestern University
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Stephanie Rangel, Research Assistant Professor of Dermatology, Northwestern University
Other Study IDs: STU00001056
Record Dates: First submitted 2016-05-04; First posted 2016-08-26 (Estimated); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Vulvar Disease; Lichen Sclerosus; Lichen Planus; Vulvodynia
MeSH Terms: conditions — Vulvar Diseases; Lichen Sclerosus et Atrophicus; Lichen Planus; Vulvodynia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women in the Vulvar Specialty Clinic: Information will be collected from all patients presenting with vulvar complaints who have been seen by Dr. Schlosser in the Vulvar Mucosal Specialty Clinic at Northwestern Medical Group.

SUMMARY:
This study aims to develop a clinical database of patients presenting with vulvar complaints in order to comprehensively assess the presentation and current trends in management of vulvar disease.

DETAILED DESCRIPTION:
Vulvar disorders are common, but their frequency and importance are often under-recognized. The spectrum of vulvar disease is vast and includes congenital malformations, inflammatory mucocutaneous diseases, blistering and erosive diseases, benign and malignant tumors, autoimmune disorders, infectious diseases, and various idiopathic conditions. Evaluation and management of genital complaints and dermatoses are complicated by the frequent multifactorial nature of vulvar symptoms and variable clinical expressions of disease on the vulva. In many cases, empiric treatment is instituted in the absence of a definitive diagnosis. Of note, expertise in the diagnosis and management of vulvar disorders is often lacking on the parts of gynecology, dermatology and primary care physicians.

The investigators seek to analyze the data on this patient population at Northwestern Memorial Hospital (NMH) and the outpatient clinics of the Northwestern Memorial Faculty Foundation (NMFF) to better define the clinical spectrum of vulvar disease. The investigators will also assess approaches to the diagnosis and management of patients with vulvar disease with attention given to clinical outcome and the impact on quality of life. This information with help the investigators to better understand the scope of care these patients currently receive, to identify deficits in current practice, and to advance potential new standards of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patients seen at Northwestern Medical Group Department of Dermatology who were seen by Dr. Bethanee Schlosser and/or other members of the Vulvar Mucosal Specialty Clinic team in any of their respective clinic settings.

Exclusion Criteria:

* Patients who refuse complete mucocutaneous examination.
* Patients who refuse recommended diagnostic procedures.
* Pregnant women or prisoners.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women seen at the Vulvar Mucosal Specialty Clinic
Sampling Method: Probability Sample
Enrollment: 719 (Actual)
Dates: Start 2016-04; Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Clinical database of patients presenting with vulvar complaints in order to comprehensively assess the presentation and current trends in the management of vulvar disease | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Potential prognostic indicators in various vulvar conditions | Through study completion, an average of 1 yea

CONTACTS AND LOCATIONS:
Overall Officials: Bethanee J Schlosser, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No